CLINICAL TRIAL: NCT05753267
Title: Clinical Study to Evaluate the Possible Efficacy of Fenofibrate in Patient With Ulcerative Colitis
Brief Title: Fenofibrate in Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Hend El-Said Abo Mansour, Faculty of Pharmacy, Menoufia University (Unknown); Monir Hussein Bahgat, Faculty of Medicine, Mansura University (Unknown)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.23
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mesalamine; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Mesalamine group will receive 1 g mesalamine three times daily for 6 months
  Interventions: Drug: Mesalamine
- Fenofibrate group (Active Comparator): Fenofibrate group will receive 1 g mesalamine three times daily plus Fenofibrate (160 mg/day) for 6 months
  Interventions: Drug: Fenofibrate 160mg

INTERVENTIONS:
Drug: Mesalamine — Mesalamine (also known as mesalamine or 5- amino salicylic acid, 5-ASA) has a well-established role in UC management. It is the first line therapy for mild to moderate UC and it is considered the cornerstone in the management of UC
  Arms: Control Group
Drug: Fenofibrate 160mg — Fibrates, which are specific pharmacological agonists of PPARα, have been widely used in the treatment of hypercholesterolemia and hypertriglyceridemia.
  Arms: Fenofibrate group

SUMMARY:
Fibrates, which are specific pharmacological agonists of PPARα, have been widely used in the treatment of hypercholesterolemia and hypertriglyceridemia. Apart from their metabolic action, anti-inflammatory properties of fibrates have been described, including inhibition of NF-kappa B signaling and pro-inflammatory cytokine production. 4 Fenofibrate, an important peroxisome proliferator-activated receptor-a (PPAR- α) agonist, is widely used in clinical as a triglyceride (TG)-lowering agent.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is an idiopathic, chronic inflammatory disease characterized by diffused inflammation of the colon and rectum mucosa, however the exact underlying mechanisms of UC remain poorly understood. UC is strongly dependent on cellular immune reaction and exaggerated inflammatory response due to genetic, immune and environmental factors.

PPARα has been proposed as a key lipid metabolism modulator and regulator of inflammation. There are three isotypes of PPAR (α, β and ȣ) which have distinct but overlapping functions.

Fibrates, which are specific pharmacological agonists of PPARα, have been widely used in the treatment for hypercholesterolemia and hypertriglyceridemia. Apart from their metabolic action, anti-inflammatory properties of fibrates have been described, including inhibition of NF-kappa B signaling and pro-inflammatory cytokine production. 4 Fenofibrate, an important peroxisome proliferator- activated receptor-a (PPAR- α) agonist, is widely used in clinical as a triglyceride (TG)-lowering agent

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both males and females will be included
* Negative pregnancy test and effective contraception.
* Mild and moderate UC patients diagnosed and confirmed by an endoscope

Exclusion Criteria:

* Breastfeeding
* Significant liver and kidney function abnormalities
* Colorectal cancer patients
* Other inflammatory bowel diseases (CD).
* Patients with severe UC
* Patients taking rectal or systemic steroids
* Patients taking immunosuppressives or biological therapies
* Addiction to alcohol and/or drugs
* Known allergy to the Fenofibrate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the change in disease activity index and the improvement in health-related quality of life (HRQL) | 6 months
  HRQL questionnaire will be assessed according to bowel symptoms, emotional symptoms, systemic symptoms, and social symptoms.

SECONDARY OUTCOMES:
The secondary endpoint is estimated by changes in serum interleukin (IL-6) and nitric oxide (NO) | 6 months
  The secondary endpoint is estimated by changes in serum interleukin (IL-6) and nitric oxide (NO)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Unuversity, Tanta, Egypt

REFERENCES:
- [Derived] Aldossary KM, Abdallah MS, Kamal N, Bahgat MM, Alrubia S, Alsegiani AS, Bahaa MM, Hassan AS, El-Khateeb E. Therapeutic Modulation of IL-6/STAT-3 and Nitric Oxide by Fenofibrate in Patients With Ulcerative Colitis: A Randomized Controlled Pilot Study. Pharmacotherapy. 2025 Dec;45(12):840-851. doi: 10.1002/phar.70088. Epub 2025 Dec 2. PMID 41330887